CLINICAL TRIAL: NCT07207200
Title: The Effects of Morning Light Therapy on IBD Activity and Symptoms
Brief Title: Impact of Morning Light Therapy in IBD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Robert Hirten, Associate Professor, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY-24-01623
Record Dates: First submitted 2025-09-03; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-10

CONDITIONS: Inflammatory Bowel Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Intervention Model Description: One hour of morning light therapy each day for four weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adult patients with Ulcerative Colitis (UC) (Experimental): Adult patients with ulcerative colitis (UC)
  Interventions: Device: Morning Light Therapy

INTERVENTIONS:
Device: Morning Light Therapy — One hour of morning light therapy each day for four weeks

SUMMARY:
The pilot study will focus on the effects of morning light therapy (MLT) in adult patients with ulcerative colitis (UC) who have evidence of poor sleep quality and active inflammation. The specific population is at risk for circadian rhythm sleep-wake disorders and has significant potential benefit from circadian realignment, which may lead to improved sleep quality and, ultimately, UC-related inflammatory activity. During an initial one-week lead-in period, participants will obtain baseline circadian-related labs, complete symptom-related surveys, and use a wearable device continuously to obtain baseline sleep-wake data. After the lead-in week, patients will undergo one hour of MLT while wearing wearable devices continuously and completing daily symptom surveys. At the end of four weeks of MLT, patients will obtain post-intervention circadian and inflammatory assessments in addition to completing the same symptom-related surveys.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ulcerative colitis and signs of inflammation (Fecal calprotectin >150 mcg/g and/or CRP >5)

Exclusion Criteria:

* Known pregnancy or currently lactating women
* Current malignancy or active treatment for previously diagnosed malignancy. Patients with squamous and basal cell cancer of the skin are eligible for the study.
* Serious co-morbidity including: Immunodeficiency, recent myocardial infarction or stroke, history of renal or hepatic failure, infection such as abscess, opportunistic infection, or sepsis.
* Patients with pacemaker or defibrillators
* The use of medications known to affect autonomic nervous system function, including but not limited to beta-blockers and benzodiazepines.
* Comprehension of the English language not adequate to understand the questionnaires
* Recent changes in IBD directed therapies within the last 3 months
* Regular use of antidiarrheal agents.
* Regular use of medications that have been shown to impair sleep (e.g. steroids, stimulants). If willing (and medically appropriate) to washout for 4 weeks, participant can be then enrolled in the study
* Regular use of sleep medications including but not limited to: benzodiazepine hypnotics, non-benzodiazepine hypnotics, antipsychotics, and melatonin. If willing (and medically appropriate) to washout for 4 weeks, participant can be then enrolled in the study
* Patients with prior colectomy or total proctocolectomy
* History of any surgery within 3 months
* Untreated Obstructive Sleep Apnea
* Blindness or severely impaired, uncorrected vision
* Employment which includes nocturnal shift work
* Traveling multiple time zones within the study time frame
* Any marijuana or illicit drugs use within one month of enrollment or ongoing basis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
C-reactive protein (CRP) level | week 4
  C-reactive protein (CRP) is produced by the liver. The CRP test is a general test to check for inflammation in the body.
Fecal Calprotectin (FCP) | week 4
  The fecal calprotectin is a stool test which measures intestinal inflammation.

SECONDARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System (PROMIS 10) | week 4
  A series of person-centered measures that evaluate and monitor physical, mental, and social health in adults.
Change in Microbiome composition | week 4
  Microbiome assessment
Change in Morning urine melatonin level | week 4
  Urine samples at the beginning and end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Hyder Said, Principal Investigator — Icahn School of Medicine at Mount Sinai; Robert Hirten, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
There is no IRB approval to share individual patient data